CLINICAL TRIAL: NCT01421264
Title: Gabapentin's Effects on Insomnia in Patients With Recent Concussion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Thomas Guttuso, Assistant Professor, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU3280611A
Record Dates: First submitted 2011-08-16; First posted 2011-08-22 (Estimated); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Insomnia
Keywords: concussion; gabapentin; neurontin; insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Brain Concussion | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gabapentin (Experimental)
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — 300mg capsules by mouth

SUMMARY:
In this open-label, pilot study the investigators will be assessing gabapentin's effects on insomnia and other concussion-related symptoms in patients with a recent concussion experiencing insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Head trauma causing concussion with either no loss of consciousness (LOC) or LOC < 30 minutes within previous 2 weeks.
2. ISS score at Baseline of > 14.
3. PCSS score at Baseline > 5.
4. If brain imaging has been checked, there was no intracerebral hemorrhage noted.
5. Glasgow Coma Scale score of 15 at Baseline.
6. Age of at least 14 years old.
7. Has not taken gabapentin or pregabalin any time since concussion and has no history of intolerance to gabapentin or pregabalin.
8. Has not taken any sleeping pills for previous 2 nights and agrees not to take any for the next 2 weeks.

Exclusion Criteria:

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index from Baseline to 1 week | 1 week

SECONDARY OUTCOMES:
Change in Post Concussion Symptom Scale score from Baseline to 1 week | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, Concussion Clinic, Buffalo, New York, United States